CLINICAL TRIAL: NCT05101902
Title: Pre-screening Study to Identify Adult Participants with Classic Congenital Adrenal Hyperplasia Due to 21-Hydroxylase Deficiency Who May Be Eligible for Treatment in the CAH-301 Trial with BBP-631, an Adeno-associated Virus (AAV) Serotype 5-Based Recombinant Vector Encoding the Human CYP21A2 Gene
Brief Title: A Study to Determine Eligibility for CAH-301 (A Study of Gene Therapy for Classic Congenital Adrenal Hyperplasia (CAH) [NCT04783181])
Status: Completed | Type: Observational
Sponsor: Adrenas Therapeutics Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CAH-300
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Congenital Adrenal Hyperplasia
Keywords: CAH
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Overall Study: Participants will undergo antibody and genetic screen, initial pre-screening, eligibility monitoring and eligibility confirmation for potential transition to the treatment trial center once a treatment assignment in the study CAH-301 becomes available. Participation in Study CAH-300 is permitted to continue until treatment assignment is available in the treatment trial or unless, during eligibility monitoring or eligibility
  Interventions: Other: Pre-Screening

INTERVENTIONS:
Other: Pre-Screening — No intervention given

SUMMARY:
This pre-screening study is designed to determine potential eligibility of adults with classic CAH due to 21-hydroxylase deficiency (21-OHD) for participation in the CAH-301 [NCT04783181] gene therapy trial with BBP-631.

DETAILED DESCRIPTION:
Adult participants diagnosed with classic CAH due to 21-OHD and who are taking glucocorticoids as treatment for CAH will undergo assessments to determine their potential eligibility for participation in the adult CAH-301 treatment trial with BBP-631.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and non-pregnant females with classic CAH (simple virilizing or salt-wasting) due to 21-OHD
* Screening/baseline 17-OHP levels > 5-10 × ULN
* Is on a daily regimen of glucocorticoid
* Naïve to prior gene therapy or AAV-mediated therapy

Exclusion Criteria:

* Positive for anti-AAV5 antibodies
* History of adrenalectomy and has no significant liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants diagnosed with classic CAH due to 21-OHD
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants Potentially Eligible for CAH-301 Study | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Science37, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Description: Adrenas Therapeutics Website — https://adrenastx.com
- See also: CAH Gene Therapy Website — https://cahgenetherapy.com